CLINICAL TRIAL: NCT02519764
Title: Evaluation of the Impact of a Hydration Protocol "at Thirst" on Natremia of the Ultra Trail du Mont-Blanc, 2015 Runners
Acronym: NATRITRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: DOKEVER (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LOCAL/2015/OM-01; 2015-A00675-44 (Other: ANSM)
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-08

CONDITIONS: Athletes; Healthy
Keywords: volunteer runners who are participating in the 2015 Mont Blanc Ultra Trail; hydration protocol; natremia; Volunteers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydration when thirsty (Experimental): Volunteers in this arm habitually follow a hydration protocol that advises hydration when thirst is felt.
  Interventions: Other: Hydration when thirsty.
- Not hydration when thirsty (Experimental): Volunteers in this arm habitually follow any other kind of hydration protocol, i.e. not a "hydration when thirsty" protocol.
  Interventions: Other: Not hydration when thirsty

INTERVENTIONS:
Other: Hydration when thirsty. — Volunteers in this arm habitually follow a hydration protocol that advises hydration when thirst is felt.
  Arms: Hydration when thirsty
Other: Not hydration when thirsty — Volunteers in this arm habitually follow any other kind of hydration protocol, i.e. not a "hydration when thirsty" protocol.
  Arms: Not hydration when thirsty

SUMMARY:
The main objective of this study is to evaluate the impact of a hydration protocol "at thirst" compared to other "not at thirst" hydration protocols on the changes in serum sodium in runners of the Ultra Trail Mont-Blanc (UTMB) in 2015.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To assess the relationship between hydration protocols and the dropout rate. B. To evaluate the correlation between body weight change before and after the race and serum sodium before and after the race.

C. To evaluate the change in serum sodium into major types of conventional hydration protocols.

D. To evaluate the incidence of adverse events (cramps, gastrointestinal symptoms, etc ...) depending on the hydration protocol and the serum sodium.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have given his/her informed and signed consent
* The subject must be insured or beneficiary of a health insurance plan
* The subject is participating in the 2015 Mont-Blanc Ultra Trail and has no contra-indication for ultra-trail activities

Exclusion Criteria:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection, under tutorship or curatorship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject is pregnant or breastfeeding

The subject will be excluded from the study in case of early drop out (before 15 km of trail).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Natremia (mmol/L) | Baseline
Natremia (mmol/L) | at finish, Days 0 to 2

SECONDARY OUTCOMES:
Weight (kg) | Baseline
Weight (kg) | at finish, Days 0 to 2
What year did you first start running regularly? | Baseline
  (pre-race questionnaire)
What year did you first start running ultra-trail races? | Baseline
  (pre-race questionnaire)
How many 100 miles or Ultra-trails races have you completed? | Baseline
  (pre-race questionnaire)
How many 100 miles or Ultra-trails races have you started but not finished? | Baseline
  (pre-race questionnaire)
What was your AVERAGE WEEKLY running training distance during the 3 months before the UTMB? | Baseline
  (pre-race questionnaire)
What was your HIGHEST running training distance IN ONE WEEK during the 3 months before the UTMB? | Baseline
  (pre-race questionnaire)
What was your LONGEST race or training run during the 3 months before the UTMB? | Baseline
  (pre-race questionnaire)
If you regularly take any medications, please list those here : | Baseline
  (pre-race questionnaire)
What were the main factors you used to decide how much to drink during the race? | Baseline
  (You may select more than one factor, but please be sure to select at least one factor.)
  Thirst(1) A pre-determined drinking schedule according to distance or time (2) The maximum amount I could tolerate (3) The amount of change in my body weight (4) My urine color (5) Other (please specify)
  (pre-race questionnaire)
What will you primarily drink during the race? | before start of race, day -1
  (Please select only one drink option.)?
  Water only (1) Mostly water and some electrolyte containing drink (2) About an equal amount of water and electrolyte containing drink (3) Mostly electrolyte containing drink and some water (4) Only electrolyte containing drink (5) Other (please specify): (6)
Indicate if you plan to use sodium supplements: yes/no | Baseline
  (pre-race questionnaire)
What is the estimated number of sodium supplements you plan to use during the race? | Baseline
  (Please only enter a number for the supplements you use. In other words, you do not need to enter a zero if you did not use the supplement.)
  Succeed S! Caps (1) Hammer Endurolyte Capsules (2) Hammer Endurolytes Fizz Tablets (3) SaltStick Caps (4) SaltStick Caps Plus (5) Nuun Electrolyte Enhanced Drink Tabs (6) GU Roctane Electrolyte Capsules (7) GU Brew Electrolyte Tablets (8) Lava Salts Capsules (9) Other (please specify) (10) Other (please specify) (10) Other (please specify) (10)
  (pre-race questionnaire)
Reflux/heartburn BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Bloating BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Stomach cramps/pain BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Nausea BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Vomiting BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal cramps/pain BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Flatulence BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Side ache/stitch BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Urge to defecate BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Loose stool/diarrhea BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal bleeding/bloody feces BEFORE THE START OF THE RACE ? | after race, days 0 to 2
  What GI symptoms did you experience… BEFORE THE START OF THE RACE ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Reflux/heartburn FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Bloating FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Stomach cramps/pain FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Nausea FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Vomiting FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal cramps/pain FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Flatulence FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Side ache/stitch FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Urge to defecate FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Loose stool/diarrhea FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal bleeding/bloody feces FROM THE START TO COURMAYEUR ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM THE START TO COURMAYEUR ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Reflux/heartburn FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Bloating FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Stomach cramps/pain FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Nausea FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Vomiting FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal cramps/pain FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Flatulence FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Side ache/stitch FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Urge to defecate FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Loose stool/diarrhea FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal bleeding/bloody feces FROM COURMAYEUR TO CHAMONIX ? | after race, days 0 to 2
  What GI symptoms did you experience… FROM COURMAYEUR TO CHAMONIX ? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Did gastrointestinal (GI) symptoms affect your race performance? yes/no | after race, days 0 to 2
  (post-race questionnaire)
Reflux/heartburn IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Bloating IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Stomach cramps/pain IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Nausea IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Vomiting IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal cramps/pain IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Flatulence IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Side ache/stitch IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Urge to defecate IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
Loose stool/diarrhea IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Intestinal bleeding/bloody feces IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? | after race, days 0 to 2
  What GI symptoms did you experience… IN THE PAST (PRIOR TO UTMB) WHILE RUNNING? Please mark the severity of each symptom using the scale of "None", "Mild", "Moderate", "Severe", or "Very Severe"
  (post-race questionnaire)
Did you use any medications (including prescription and over-the-counter) immediately before or during the 2015 UTMB? (post-race questionnaire) | after race, days 0 to 2
  If so, please list
Did you have any muscle cramps during the 2015 UTMB? | after race, days 0 to 2
  Yes Almost, but was able to control any full-blown cramping No
  (post-race questionnaire)
If yes, In which muscles did you have an issue with cramping during the 2015 UTMB? | after race, days 0 to 2
  Calf muscles Quadriceps Hamstrings Hip flexors (muscles in front of pelvis and top of leg) Other(s) (please specify): ____________________
  (post-race questionnaire)
If yes, Indicate which race section(s) you had issues with muscle cramps (post-race questionnaire) | after race, days 0 to 2
  Start to Courmayeur Courmayeur to Chamonix
  (post-race questionnaire)
Have you had muscle cramps during prior ultra-trail runs? yes/no | after race, days 0 to 2
  (post-race questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marès, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Nice - Hôpital St-Roch, Nice
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Mouzat K, Raoul C, Polge A, Kantar J, Camu W, Lumbroso S. Liver X receptors: from cholesterol regulation to neuroprotection-a new barrier against neurodegeneration in amyotrophic lateral sclerosis? Cell Mol Life Sci. 2016 Oct;73(20):3801-8. doi: 10.1007/s00018-016-2330-y. Epub 2016 Aug 10. PMID 27510420